CLINICAL TRIAL: NCT04228991
Title: Randomized Trial of Hypofractionated LocoRegional Radiotherapy in Breast Cancer and Lymphedema (RHEAL)
Brief Title: Hypofractionated LocoRegional Radiotherapy in Breast Cancer
Acronym: RHEAL
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ontario Clinical Oncology Group (OCOG) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OCOG-2019-RHEAL
Record Dates: First submitted 2020-01-09; First posted 2020-01-14 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-07

CONDITIONS: Breast Neoplasms; Radiotherapy; Lymphedema
Keywords: Hypofractionated; Locoregional; Breast Cancer; Lymphedema
MeSH Terms: conditions — Breast Neoplasms; Lymphedema

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Conventional fractionation for locoregional radiotherapy
  Interventions: Radiation: Locoregional radiation treatment - Conventional fractionation
- Experimental (Experimental): Hypofractionation for locoregional radiotherapy
  Interventions: Radiation: Locoregional radiation treatment - Hypofractionation

INTERVENTIONS:
Radiation: Locoregional radiation treatment - Conventional fractionation — 40 Gray in 15 daily fractions over 3 weeks
  Arms: Control
Radiation: Locoregional radiation treatment - Hypofractionation — 26 Gray in 5 daily fractions over 1 week
  Arms: Experimental

SUMMARY:
The primary objective of this study is to determine if hypofractionated RT delivered over 1 week to the breast or chest wall and regional nodes (26Gy in 5 daily fractions) following BCS or mastectomy, is non-inferior to conventional fractionation to the breast or chest wall and regional nodes delivered over 3 weeks (40Gy in 15 daily fractions) in patients with node-positive breast cancer.

DETAILED DESCRIPTION:
A multi-centre, randomized, non-inferior, phase III study comparing two radiation treatment modalities, conventional fractionation with hypofractionation for locoregional RT. Eligible, consenting patients with newly diagnosed and histologically confirmed invasive carcinoma of the breast without evidence of metastatic disease; treated with definitive surgery [BCS or mastectomy with nodal staging using sentinel lymph node biopsy (SLNB) or axillary lymph node dissection (ALND)] will be randomized in a 1:1 fashion to either conventional locoregional RT (control group) or hypofractionated locoregional RT (experimental group). Stratification factors include: body mass index, the performance of ALND, type of surgery (BCS or mastectomy) and clinical centre.

Study participants will be assessed for lymphedema, the primary outcome, by measuring arm volume. Arm mobility will be assessed by measuring arm movement. Study participants will be assessed for acute and late radiation toxicities, during and post RT. Study participants will be followed and assessed annually for breast cancer recurrence (BCR), new second cancers, quality of life (QOL) and overall survival. Cost effectiveness and cost utility will also be determined. The planned sample size is 588 study participants. The study will be conducted at clinical centres throughout Canada.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed invasive carcinoma of the breast.
2. Treated with definitive surgery (BCS or mastectomy with nodal staging using SLNB or ALND) with clear margins of excision.* Note: *Patients with limited positive posterior margin where disease is resected to chest wall or limited positive anterior margin where disease is resected to dermis are eligible.
3. Candidate for locoregional radiotherapy: breast cancer stage after definitive surgery:

   * Neoadjuvant chemotherapy was not administered: pathologic stage T3N0,T1-3 N1-2**

     ** patients with nodal micromets (N1mi) are eligible
   * Neoadjuvant chemotherapy was administered: clinical stage T3N0, T1-3, N1-2 and pathologic stage T0-3, N0-2†

     * Patients who are clinically N1-2 prior to chemotherapy should be confirmed histologically unless it is clear that they are node positive. Patients who are deemed node negative prior to chemotherapy but are node positive following chemotherapy are eligible. Patients who are node positive prior to chemotherapy and who have complete response in the lymph nodes are also eligible.
4. No evidence of metastatic disease.

Exclusion Criteria:

1. Age < 18 years.
2. Clinical stages T4 and/or N3.
3. Clinical lymphedema in the ipsilateral arm or breast/chest wall.
4. Any prior history, not including index cancer, of ipsilateral invasive breast cancer or ipsilateral DCIS treated with radiation therapy. (Patients with previous ipsilateral DCIS or LCIS not treated with radiation are eligible.)
5. Synchronous or previous contralateral breast cancer.(Patients with previous contralateral DCIS or LCIS not treated with radiation are eligible.)
6. History of non-breast malignancy within the last 5 years other than non-melanoma skin cancer or treated in-situ carcinoma.
7. Neoadjuvant endocrine therapy. (Extended neoadjuvant endocrine therapy is not permitted. Endocrine therapy exposure for 12 weeks or less prior to surgery is acceptable.)
8. Breast reconstruction.
9. Presence of known medical conditions that would preclude follow-up for 5 years.
10. Previous radiotherapy to the ipsilateral breast or chest wall or serious non-malignant disease e.g. scleroderma, severe lung or heart disease that would preclude radiotherapy.
11. Known pregnancy or currently lactating.
12. Geographic inaccessibility for follow-up.
13. Inability to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 588 (Estimated)
Dates: Start 2021-02-10 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Lymphedema | 3 years post randomization
  Lymphedema defined as relative volume change (RVC) ≥10%

SECONDARY OUTCOMES:
Breast cancer recurrence | Annually for 5 years post randomization
  Both locoregional and distant recurrence and second cancers
Mortality | Annually for 5 years post randomization
  Survival
Radiation toxicity | During last week of radiotherapy, at 3 months post radiotherapy and annually for 5 years post randomization
  Acute and late radiation toxicity
Arm mobility | 1 and 3 years post randomization
  Assessed by measuring the straight lateral abduction of both the ipsilateral and contralateral arm
Patient Quality of Life with respect to daily health and activities | During last week of radiotherapy, at 3 months post radiotherapy and 1 and 3 years post randomization
  Impact on quality of life will be assessed with the European Organization for Research in Treatment of Cancer and the Breast Cancer Specific Module 23. The scale is 1 to 4 where a higher score means a worse outcome.
Perception of lymphedema | During last week of radiotherapy, at 3 months post radiotherapy and 1 and 3 years post randomization
  Impact of lymphedema on quality of life will be assessed with the National Surgical Adjuvant Breast and Bowel Project questionnaire. The scale is 1 to 5 where a higher score means a worse outcome.
Perception of breast cosmesis | 1 and 3 years post randomization
  Patient-reported breast cosmesis using a Breast Cosmesis Questionnaire to study the late effects of radiation.
Health Care Resource Utilization | During radiotherapy, at 3 months post radiotherapy and annually for 5 years post randomization
  Health Care Resource Utilization will be estimated using dates and duration of radiotherapy treatment and emergency department visits and hospitalizations.
Patient Costs | During last week of radiotherapy, at 3 months post radiotherapy and 1 and 3 years post randomization
  Patient costs will be assessed using a Time Off Work Questionnaire to study the financial impact of breast cancer and its treatment

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Whelan, MD, Principal Investigator — Juravinski Cancer Centre, McMaster University, Hamilton
Locations (20):
- Canada (20):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - BC Cancer - Centre for the Southern Interior, Kelowna, British Columbia
  - BC Cancer - Centre for the North, Prince George, British Columbia
  - BC Cancer - Vancouver Centre, Vancouver, British Columbia
  - BC Cancer - Vancouver Island Centre, Victoria, British Columbia
  - Northeast Cancer Centre, Health Sciences North, Greater Sudbury, Ontario
  - Juravinski Cancer Centre, Hamilton, Ontario
  - London Regional Cancer Program, London, Ontario
  - The Ottawa Hospital Regional Cancer Centre, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre - Odette Cancer Centre, Toronto, Ontario
  - Princess Margaret Cancer Centre - UHN, Toronto, Ontario
  - Hotel-Dieu de Lévis (CISSS CA), Lévis, Quebec
  - CIUSSS de l'Est-de-l'Île de Montréal, Hôpital, Maisonneuve-Rosemont, Montreal, Quebec
  - McGill University Health Centre-Cedars Cancer Centre, Montreal, Quebec
  - CHUM - Centre Hospitalier de L'Universite de Montreal, Montreal, Quebec
  - CHU-de Québec-Université de Laval, Québec, Quebec
  - Sherbrooke University Hospital Centre, Sherbrooke, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan